CLINICAL TRIAL: NCT04975789
Title: Information Visualization to Improve Pain Communication Between Providers, Interpreters, and Patients With Limited English Proficiency
Brief Title: Visualizations to Improve Pain Communication Between Patients, Interpreters, and Providers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-1256; A545000 (Other: UW Madison); NUR/FACULTY AFFAIRS/ADMIN (Other: UW Madison); Protocol Approved 10/11/21 (Other: UW Madison); 1K23NR019289-01A1 (NIH)
Record Dates: First submitted 2021-07-14; First posted 2021-07-23 (Actual); Results first posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Communication; Pain
Keywords: pain assessment; limited English proficiency; mutual understanding
MeSH Terms: conditions — Communication; Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care Control (No Intervention): Standard of Care
- InfoViz Intervention (Experimental): Pain information visualization (InfoViz) tool, Trained interpreters will use the InfoViz tool twice, before and during the clinical encounter
  Interventions: Other: InfoViz

INTERVENTIONS:
Other: InfoViz — The pain InfoViz tool is a two-page paper tool that consists of an explanation of how to use the tool in both Hmong and English, a culturally-appropriate Faces pain severity scale, pain body diagram, and 13 pain qualities in the form of icons representing each pain quality metaphor. The interpreter explains the instructions in Hmong, then marks the body areas corresponding to the location of pain reported by the participant, and marks the pain qualities expressed by the metaphors selected by the Hmong patient. In the clinic appointment, the interpreter communicates to the physician, in English, the pain location and qualities identified by the participant, using the medical terms identified on the InfoViz tool.
  Other Names: Pain Assessment Tool
  Arms: InfoViz Intervention

SUMMARY:
The purpose of this study is to pilot test a pain assessment information visualization (InfoViz) tool to facilitate communication about pain severity, location, and quality to increase mutual understanding between patients with limited English proficiency (LEP), interpreters, and providers during pain assessment. 40 participants will be enrolled and can expect to be on study for up to 4 weeks.

DETAILED DESCRIPTION:
The purpose of this study is to pilot test a pain assessment information visualization (InfoViz) tool to facilitate communication about pain severity, location, and quality to increase mutual understanding between patients with limited English proficiency (LEP), interpreters, and providers during pain assessment.

The investigators focus on the LEP Hmong because pain is particularly problematic for this group. The Hmong describe pain using visual metaphors that are inconsistent with providers' knowledge and interpreters struggle to translate metaphors accurately between patients and providers. The goals of the study are (1) to examine the feasibility of implementing the pain InfoViz tool, (2) to explore congruency of patient-interpreter-provider triads' mutual understanding (MU) of pain severity, location, and quality, and (3) to evaluate outcome measures selected to capture satisfaction with communication, pain relief, and pain interference with life and explore variables identified in the InfoViz tool conceptual framework (MU of pain assessment information, satisfaction with communication, pain diagnosis and treatment).

The investigators will first collect data from 20 participants under the usual care control condition (i.e., interpreters verbally interpreting and communicating pain descriptions), followed by data collection from another 20 participants under the intervention condition (i.e., interpreters using verbal descriptions and the InfoViz tool).

The investigators believe that the pain assessment InfoViz tool will increase mutual understanding of pain severity, location, and quality between patients, interpreters, and providers, and consequently lead to increased satisfaction with communication, greater pain relief and reduced pain interference with daily life through better-informed diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

* age 18 and up
* Hmong patients that indicate they do not speak English well (LEP)
* self reported pain

Exclusion Criteria:

* indicate that they speak English well

Interpreter Inclusion Criteria:

* 13 years old or greater
* self-identify as interpreting for a Hmong individual in the health care setting

Interpreter Exclusion Criteria:

* telephone interpreters as they are unable to view and use the InfoViz tool

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2021-10-07 (Actual); Primary Completion 2023-01-06 (Actual); Study Completion 2023-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maichou Lor, PhD, RN, Principal Investigator — University of Wisconsin, Madison
Locations (2):
- United States (2):
  - Access Community Health Center, Madison, Wisconsin
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lor M, Li A, Brown R, Swedlund MP, Hawkins JG, Nolander ET, Chewning B. Improving pain communication between limited English-speaking Hmong patients, medical interpreters, and health care providers in primary care: A pilot study. Res Nurs Health. 2024 Jun;47(3):289-301. doi: 10.1002/nur.22363. Epub 2024 Jan 4. PMID 38175545

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from October 2021 to February 2023.
Pre-assignment Details: Enrolled participants have an associated participant group, which includes the patient, the interpreter, and the provider.
Groups:
- Usual Care: Use interpreter but no pain information visualization tool used
- Interpreters: People able to speak both English and Hmong, part of the participant triad of with Patient, Interpreter, Provider.
- Providers: Providers who completed surveys, part of the participant triad of with Patient, Interpreter, Provider.
Period: Overall Study
Arm/Group | Usual Care | InfoViz Intervention | Interpreters | Providers
Started | 18 | 18 | 4 (4 unique interpreters were part of 36 separate patient, interpreter, provider triads.) | 21 (21 unique providers returned surveys)
Completed Follow Up | 15 | 13 | 4 | 21
Completed | 18 | 18 | 4 | 21
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Interpreters: People who speak English and Hmong, part of the Patient, Interpreter, Provider triad.
- Providers: Providers who returned surveys, part of the Patient, Interpreter, Provider triad.
- Total: Total of all reporting groups
Arm/Group | Usual Care | InfoViz Intervention | Interpreters | Providers | Total
Number analyzed (Participants) | 18 | 18 | 4 | 21 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] — The total mean age reported is for the 36 patients involved in the study and excludes the mean age of interpreters and providers.
  years | 56 (12.43) | 57 (11.82) | 36 (10.78) | 41.24 (11.33) | 56 (11.98)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 14 | 15 | 1 | 15 | 45
  Male | 4 | 3 | 3 | 5 | 15
  Unknown - Did Not Report | 0 | 0 | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 18 | 18 | 4 | 20 | 60
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 18 | 18 | 4 | 2 | 42
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 19 | 19
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 18 | 4 | 21 | 36

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Eligible Patients Enrolled
Description: Feasibility with respect to recruitment will be measured by the percent of eligible patients who enroll.
Time Frame: up to 1 day
Measure: Count of Participants; unit: Participants
Groups:
- InfoViz: Pain information visualization (InfoViz) tool, Trained interpreters will use the InfoViz tool twice, before and during the clinical encounter
Arm/Group | Usual Care | InfoViz
Number analyzed (Participants) | 18 | 18
Participants | 18 | 18

2. Primary Outcome: Proportion of Patients Who Complete the Study
Description: Feasibility with respect to retention will be measured by the proportion of patients who complete the study.
Time Frame: up to 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | InfoViz Intervention
Number analyzed (Participants) | 18 | 18
Participants | 18 | 18

3. Primary Outcome: Percentage of InfoViz Tools Completely Filled Out
Description: Feasibility with respect to tool use will be measured as the proportion of InfoViz tools with pain severity marked, at least one pain location marked, and at least one pain quality marked on the InfoViz tool.
Time Frame: up to 1 day
Population: Enrolled patients have an associated participant group (a triad), which includes the patient, the interpreter, and the provider.
Measure: Number; unit: percentage of InfoViz tool
Units Other Than Participants: InfoViz Tools
Arm/Group | InfoViz Intervention
Number analyzed (Participants) | 18
Number analyzed (InfoViz Tools) | 18
percentage of InfoViz tool | 100

4. Primary Outcome: Percentage of Items Correctly Performed on the Investigator Designed Fidelity Checklist
Description: Feasibility will be in part measured by InfoViz tool fidelity. The percentage of items correctly performed by participants on the investigator-designed fidelity checklist will be reported.
Time Frame: up to 1 day
Population: This outcome is informed by the interpreter in the participant triad.
Measure: Mean (Standard Deviation); unit: percent of checklist items
Units Other Than Participants: checklist items
Arm/Group | InfoViz Intervention
Number analyzed (Participants) | 18
Number analyzed (checklist items) | 18
percent of checklist items | 83 (10)

5. Primary Outcome: Percentage of Congruency in Mutual Understanding: Patient to Interpreter
Description: One question item from the 6-item Mutual Understanding Scale (MUS) asks participants about their main symptom (i.e., "What was the most important health complaint for which the physician was visited?") and providers to report participants' main symptom (e.g., "What was the most important health complaint for which the patient consulted with you?"). The percentage of congruency between the patient and interpreter response, from 0-100 where 100 is total congruency.
Time Frame: up to 1 day
Population: Enrolled participants have an associated participant group, which includes the patient, the interpreter, and the provider.
Measure: Number; unit: percentage of total congruency
Arm/Group | Usual Care | InfoViz Intervention
Number analyzed (Participants) | 18 | 18
percentage of total congruency
  Pain Location | 20 | 22
  Pain Quality | 20 | 11
  Pain Severity | 30 | 28

6. Secondary Outcome: Participant Satisfaction With Communication Answer
Description: Satisfaction with communication will be measured using one item, "Overall, how satisfied are you with your doctor's communication with you about pain?" with response categories of very satisfied, satisfied, neither satisfied nor dissatisfied, dissatisfied, or very dissatisfied. Mean score between 1-5, where 5 indicate higher satisfaction and 1 indicate very dissatisfaction, was calculated across participant groups (i.e., patient, interpreter, provider).
Time Frame: up to 1 day
Population: Enrolled participants have an associated participant group, which includes the patient, the interpreter, and the provider (18 participant triads). Each group member are surveyed for satisfaction.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | InfoViz Intervention
Number analyzed (Participants) | 38 | 37
score on a scale
  Patient: number analyzed (Participants) | 18 | 18
  Patient | 3.21 (0.78) | 3.44 (0.61)
  Interpreter: number analyzed (Participants) | 4 | 4
  Interpreter | 4.33 (0.59) | 4.55 (0.51)
  Provider: number analyzed (Participants) | 16 | 15
  Provider | 4.2 (0.51) | 4.6 (0.63)

7. Secondary Outcome: Participant Pain Relief Measured Using a 5 Point Verbal Rating Scale
Description: Participants will be asked to rate the amount of pain relief experienced since the clinic visit using a 5-point Verbal Rating Scale: none, slight, moderate, lots, complete. A mean score between 1-5, where higher scores equal complete pain relief.
Time Frame: one time post 4-6 weeks after the clinic vist
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | InfoViz Intervention
Number analyzed (Participants) | 18 | 18
score on a scale | 1.6 (0.99) | 1.88 (1.21)

8. Secondary Outcome: Participant Response to Pain Interference Question
Description: One question item derived from the 12-Item Short-Form Health Survey, "During the past 4 weeks, how much did pain interfere with your normal work including both work outside the home and housework?" with response options: "not at all," "a little bit," "moderately," "quite a bit," or "extremely." The number of participants who responded to each condition will be reported. Mean score 1-5, where higher score indicates extreme pain interference, was calculated.
Time Frame: usual care participants assessed at baseline and InfoViz participants assessed at 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | InfoViz Intervention
Number analyzed (Participants) | 18 | 18
score on a scale | 1.6 (0.99) | 1.84 (1.21)

9. Secondary Outcome: Quality of Communication Answer
Description: Quality of communication will be measured using one item, "Overall, how would you rate this doctor's communication about pain with you? " with response items of excellent, very good, good, fair, or poor. Mean scores of 1 to 5, where higher number indicates excellent quality of communication, was calculated.
Time Frame: up to 1 day
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | InfoViz Intervention
Number analyzed (Participants) | 38 | 37
score on a scale
  Patient: number analyzed (Participants) | 18 | 18
  Patient | 3.68 (0.58) | 4.11 (0.67)
  Interpreter: number analyzed (Participants) | 4 | 4
  Interpreter | 3.50 (0.85) | 3.61 (0.97)
  Provider: number analyzed (Participants) | 16 | 15
  Provider | 3.58 (0.87) | 3.46 (0.99)

10. Primary Outcome: Percentage of Congruency in Mutual Understanding: Interpreter to Provider
Description: One question item from the 6-item Mutual Understanding Scale (MUS) asks participants about their main symptom (i.e., "What was the most important health complaint for which the physician was visited?") and providers to report participants' main symptom (e.g., "What was the most important health complaint for which the patient consulted with you?"). The percentage of congruency between the interpreter and provider, from 0-100 where 100 is total congruency.
Time Frame: up to 1 day
Population: as for outcome 5
Measure: Number; unit: percentage of total congruency
Arm/Group | Usual Care | InfoViz Intervention
Number analyzed (Participants) | 18 | 18
percentage of total congruency
  Pain Location | 90 | 56
  Pain Quality | 30 | 39
  Pain Severity | 40 | 39

11. Primary Outcome: Percentage of Congruency in Mutual Understanding: Patient to Provider
Description: One question item from the 6-item Mutual Understanding Scale (MUS) asks participants about their main symptom (i.e., "What was the most important health complaint for which the physician was visited?") and providers to report participants' main symptom (e.g., "What was the most important health complaint for which the patient consulted with you?"). The percentage of congruency between patient and provider, from 0-100 where 100 is total congruency.
Time Frame: up to 1 day
Population: as for outcome 5
Measure: Number; unit: percentage of total congruency
Arm/Group | Usual Care | InfoViz Intervention
Number analyzed (Participants) | 18 | 18
percentage of total congruency
  Pain Location | 90 | 72
  Pain Quality | 50 | 50
  Pain Severity | 20 | 50

ADVERSE EVENTS:
Description: adverse were were not monitored/assessed
Arm/Group | Usual Care | InfoViz Intervention
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-09-18): https://cdn.clinicaltrials.gov/large-docs/89/NCT04975789/Prot_000.pdf
  • Informed Consent Form (2021-12-10): https://cdn.clinicaltrials.gov/large-docs/89/NCT04975789/ICF_001.pdf